CLINICAL TRIAL: NCT00005615
Title: The Florida Melanoma Trial: A Phase I/II Trial of Post-Operative Adjuvant Radiotherapy With Concurrent Interferon-Alfa in the Treatment of Advanced Stage III Melanoma: Study Site & Coordinating Center
Brief Title: Post-Operative Adjuvant Radiotherapy With Concurrent Interferon-Alfa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11543; NCI-G00-1750 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2004-04-02 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon Alfa Plus Radiation (Experimental): Combined Therapy: interferon alfa plus radiation therapy.
  Patients receive interferon alfa IV over 20 minutes daily for 5 consecutive days a week for 4 weeks. Patients then receive radiotherapy on days 2 and 4 and interferon alfa subcutaneously (SQ) on days 1, 3, and 5 for 2.5 weeks. Interferon alfa SQ continues 3 times a week for 10 months in the absence of disease progression or unacceptable toxicity. Patients are followed every month for 3 months, then every 3 months for 2 years, then every six months until year 5, and then annually thereafter.
  Interventions: Biological: Interferon alfa; Radiation: Radiation therapy

INTERVENTIONS:
Biological: Interferon alfa — Interferon alfa as outlined in treatment arm.
Radiation: Radiation therapy — Radiation therapy as outlined in treatment arm.

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining interferon alfa plus radiation therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of interferon alfa plus radiation therapy in treating patients who have stage III or recurrent melanoma that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness and toxicity of adjuvant radiotherapy given concurrently with interferon alfa to patients with stage III or recurrent melanoma.

OUTLINE: This is a multicenter study. Patients receive interferon alfa IV over 20 minutes daily for 5 consecutive days a week for 4 weeks. Patients then receive radiotherapy on days 2 and 4 and interferon alfa subcutaneously (SQ) on days 1, 3, and 5 for 2.5 weeks. Interferon alfa SQ continues 3 times a week for 10 months in the absence of disease progression or unacceptable toxicity. Patients are followed every month for 3 months, then every 3 months for 2 years, then every six months until year 5, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 2.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primary melanoma with extensive regional node metastases (T1-4, N1, M0) OR Primary melanoma with clinically apparent metastases confirmed by lymphadenectomy (T1-4, N1-2, M0) OR Clinically detected relapse of melanoma in regional node basin, confirmed by lymphadenectomy after prior management of primary site (T1-4, N1-2, M0) OR Recurrence of melanoma in a nodal basin previously resected OR Nodal metastatic melanoma arising from unknown primary, confirmed by lymphadenectomy (Tx, N1-2, M0) Adenopathy from neck, axilla, or groin basins must meet one of the following criteria: At least 4 positive nodes containing tumor Nodal metastases at least 3 cm in size Gross extracapsular extension of tumor Recurrence after prior lymphadenectomy Completely resected disease No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 6 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 125,000/mm3 Hematocrit at least 33% Hepatic: AST, LDH, alkaline phosphatase and bilirubin no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.8 mg/dL BUN no greater than 33 mg/dL Cardiovascular: No congestive heart failure (New York Heart Association class III or IV heart disease) Neurologic: No prior CNS demyelinating or inflammatory disease No prior hereditary or acquired peripheral neuropathy No organic brain syndrome, significant impairment of cognitive function, or psychiatric disorder that would preclude study Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 18 months after study No hypersensitivity to interferon alfa or any component of the injection No history of diabetes mellitus prone to ketoacidosis No uncontrolled thyroid abnormalities No clinically significant retinal abnormalities No other significant medical or surgical condition that would preclude study No prior invasive melanoma No other prior or concurrent malignancies within the past 5 years except any in situ cancer, atypical melanocytic hyperplasia, or basal or squamous skin cancer No autoimmune disorders or immunosuppressive conditions

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior vaccine therapy allowed No prior immunotherapy, interferon, interleukins, levamisole, or other biologic response modifiers Chemotherapy: No prior chemotherapy, including infusion or perfusion therapy Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: No prior radiotherapy to the proposed site(s) of study Surgery: See Disease Characteristics Other: No other medication or treatment regimen that would preclude study No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1997-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Study Duration: 7 years
  Objective response rate according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Study Duration: 7 years
  Review of adverse events utilizing Common Toxicity Criteria (CTC) V3.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C. DeConti, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida